CLINICAL TRIAL: NCT05159843
Title: Effects of Nursing Diabetes Self-management Education on Glycemic Control and Self-care
Brief Title: Effects of Nursing Diabetes Self-management Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Rocío Romero Castillo, Principal Investigator, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Tesis-ETD-2021
Record Dates: First submitted 2021-11-22; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus, Type 1; Health Behavior
Keywords: Type 1 Diabetes; Health Education; Nurses; Self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Health Behavior; Health Education

STUDY DESIGN:
Intervention Model Description: A two-group randomized controlled trial will be used in this project. Participants in the experimental group will undergo four-session health education program, while the participants in the control group will receive the existing standard care provided by the hospital. Measurements will be conducted at the baseline prior to the intervention and at 1 an 3 months from the intervention.
Who Masked: Participant, Care Provider
Masking Description: To achieve a well balance in the randomization procedure block randomization of size 10 (with five experimental and five control) in seal envelops will be used. It will use the computerized randomization programme to generate the randomization programme to generate the randomization list using with block size of 10. A team member who will not be involved in recruitment and data collection will prepare the sealed envelopes according to the generated randomization list. After a patient is registered, a unique patient ID will be assigned to the patient based on the sequence of his/her enrolment. The envelope according to the patient's ID will be opened on site and the patient will be allocated into either one of the two groups based on the randomization list the treatment indicated.
  Both patient and nurses offering therapeutic education will be blinded in this study and they will not know the objectives of the investigation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Self-Management education (Experimental): Participants randomized to this arm receive therapeutic education during four sessions of four consecutive days. An advanced practice nurse who specializes in diabetes will teach these sessions. The sessions will have small groups of five patients and it will last of one hour each day. The outline of the session is as follow (Figure 1):
  First session: Insulin administration and blood glucose self-analysis Second session: Management of hypoglycemia and hyperglycemia Third session: Healthy diet adapted to the diabetic patient Four session: Physical exercise
  Interventions: Behavioral: Therapeutic education
- Usual care (Experimental): Participants in control group receive usual services offered in University Hospital and other local health systems for patients with diabetes, which include regular visits with a diabetes provider (primary care or endocrine) and standard Spanish Diabetes Society information pamphlets. Consultation care is centralized in the pharmacological treatment regimen, dosage and guidelines.
  Interventions: Behavioral: Therapeutic education

INTERVENTIONS:
Behavioral: Therapeutic education — Participants randomized to this arm receive therapeutic education during four sessions of four consecutive days. An advanced practice nurse who specializes in diabetes will teach these sessions. The sessions will have small groups of five patients and it will last of one hour each day. The outline of the session is as follow (Figure 1):
  First session: Insulin administration and blood glucose self-analysis Second session: Management of hypoglycemia and hyperglycemia Third session: Healthy diet adapted to the diabetic patient Four session: Physical exercise

SUMMARY:
A study protocol for analyze the influence of therapeutic education on the metabolic control of patients with type I diabetes. To measure the change in glucose levels, it will use the continuous glucose monitoring sensor that the patients have implanted. It will perform a data download prior and after to the educational intervention. An assessment of acquired knowledge will also be performed and it will be analyzed whether learning about their disease and self-care helps to improve their emotional state.

The intervention of this study is only training with therapeutic education, it does not require any type of extra test or medical or pharmacological product. It will only be necessary to answer attitudinal questionnaires by the patient

DETAILED DESCRIPTION:
A two-group randomized controlled trial will be used in this project. Participants in the experimental group will undergo four-session health education program, while the participants in the control group will receive the existing standard care provided by the hospital. Measurements will be conducted at the baseline prior to the intervention and at 1 an 3 months from the intervention.

To achieve a well balance in the randomization procedure block randomization of size 10 (with five experimental and five control) in seal envelops will be used. It will use the computerized randomization programme to generate the randomization programme to generate the randomization list using with block size of 10. A team member who will not be involved in recruitment and data collection will prepare the sealed envelopes according to the generated randomization list. After a patient is registered, a unique patient ID will be assigned to the patient based on the sequence of his/her enrolment. The envelope according to the patient's ID will be opened on site and the patient will be allocated into either one of the two groups based on the randomization list the treatment indicated.

Participants in control group receive usual services offered in University Hospital and other local health systems for patients with diabetes, which include regular visits with a diabetes provider (primary care or endocrine) and standard Spanish Diabetes Society information pamphlets. Consultation care is centralized in the pharmacological treatment regimen, dosage and guidelines.

Participants randomized to this arm receive therapeutic education during four sessions of four consecutive days. An advanced practice nurse who specializes in diabetes will teach these sessions. The sessions will have small groups of five patients and it will last of one hour each day. The outline of the session is as follow (Figure 1):

First session: Insulin administration and blood glucose self-analysis Second session: Management of hypoglycemia and hyperglycemia Third session: Healthy diet adapted to the diabetic patient Four session: Physical exercise

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of type 1 diabetes
* 18 years old and above
* Able to speak, read and listen Spanish

Exclusion Criteria:

* Have suffered from severe complications such as severe stroke, visual impairment or renal failure that interfere from severe complications such as severe stroke, visual impairment or renal failure that interfere with self-care activities
* Have a history of major psychiatric conditions (for example schizophrenia), other than depression or anxiety
* Have reading and hearing diffuculties
* Be in police custody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge in diabetes management | 3 months
  Measure by pre-test and post-test

SECONDARY OUTCOMES:
Glycemic control | 3 months
  Data obtained by the continuous glucose monitoring sensor
Healthy diet and physical exercise | 3 months
  Diabetes Self-Care Activities measure. The minimum value of this scale is 0 and the maximum is 49 points. Higher scores indicate better diabetes self-care outcomes.
Mood of patient | 3 months
  Measure by Goldberg Anxiety and Depression Scale. The minimum value of this scale is 0 and the maximum is 18 points. Higher values indicate higher levels of anxiety and depression, and therefore worse health outcomes

IPD SHARING:
Plan to Share IPD: No
According to the ethics committee and to respect data protection, clinical data will not be uploaded.
  If others researchers wants more information, they will contact the IP (Rocío Romero Castillo)

REFERENCES:
- [Derived] Romero-Castillo R, Pabon-Carrasco M, Kaknani-Uttumchandani S, Ponce-Blandon JA. Effects of Continuous Glucose Monitoring on Glycemic Control, Mental Health and Self-Management in Adults with Type 1 Diabetes: A Randomized Controlled Trial. Healthcare (Basel). 2025 Dec 5;13(24):3197. doi: 10.3390/healthcare13243197. PMID 41464266